CLINICAL TRIAL: NCT00296452
Title: The Effect of an Enhanced Nutritional Supplement on Head and Neck Cancer Patients
Brief Title: Effect of a Nutritional Supplement on H&N Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Edward Hines Jr. VA Hospital (U.S. Federal Agency)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 0033
Record Dates: First submitted 2006-02-23; First posted 2006-02-27 (Estimated); Last update posted 2006-02-27 (Estimated); Status verified 2006-02

CONDITIONS: Head and Neck Cancer
Keywords: cancer; nutrition
MeSH Terms: conditions — Head and Neck Neoplasms; Neoplasms

INTERVENTIONS:
Behavioral: behavior

SUMMARY:
To determine if using a nutritionally enhanced supplement will improve mucositis in head and neck cancer patients

DETAILED DESCRIPTION:
H&N cancer patients will be randomized to receive either a nutritionally enhanced product or standard treatment. The patients in both groups will receive nutritional counseling weekly by the RD. Anthropometric measures, available lab values, mucositis grade, and quality of life measures will be compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* Head and neck cancer 1st.2nd wk Rx read &wrte eng

Exclusion Criteria:

* receiving hospice impaired cognition

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2006-02; Study Completion 2006-02

PRIMARY OUTCOMES:
severity of mucositis

SECONDARY OUTCOMES:
weight loss, quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Foley, MS, Principal Investigator — Hines VA Hosptial; carol bier-laning, MD, Principal Investigator — Hines VA Hospital
Locations (2):
- United States (2):
  - Edward Hines, Jr. VA Hospital, Hines, Illinois
  - Hines VA Hospital, Hines, Illinois